CLINICAL TRIAL: NCT07053397
Title: A Comparative Study on the Analgesic Efficacy of Ultrasound-Guided Continuous Catheter-Based Deep Serratus Anterior Plane Block Versus Single-Injection Deep Serratus Anterior Plane Block in Patients Undergoing Breast Surgery
Brief Title: We Have Two Groups. Both Groups Received a Deep Serratus Anterior Plane Block. One Group Had a Catheter for Continuous Infusion, While the Other Received IV Analgesics Postoperatively. Analgesic Effects Between the Two Groups Were Compared
Acronym: DSAPB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medeniyet University (Other)
Responsible Party: Principal Investigator, Alper Ağbulak, Research Assistant, Istanbul Medeniyet University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: SAP001
Record Dates: First submitted 2025-06-27; First posted 2025-07-08 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Pain Management After Surgery; Regional Anaesthesia
Keywords: SAP; Deep SAP Block; Regional block; Peripheral block; Peripheral block cathather; continuous infusion via peripheral block cathather
MeSH Terms: interventions — Saposins; Population Groups

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SAPB (Active Comparator): The SAPB arm receives single shot deep serratus anterior plane block before surgery. Also receives iv analgesic treatment after post-operative duration.
  Interventions: Procedure: Serratus Anterior Plane Block (SAPB) group
- DSAPB (Experimental): The DSAPB arm receives deep serratus anterior plane block and cathather replacement before surgery. After surgery, the arm takes continous analgesic treatment via periferic block cathather.
  Interventions: Procedure: Serratus Anterior Plane Block (SAPB) group; Procedure: DSAPB

INTERVENTIONS:
Procedure: Serratus Anterior Plane Block (SAPB) group — The SAP block, which is among the chest wall blocks, provides its effect by blocking the lateral cutaneous branches of the T2-T9 intercostal nerves, n. intercostobrachial , n. longus thoracicus , n. thoracodorsal.
  SAP block can be performed in two ways: superficial and deep. The deep SAP block is administered between the serratus anterior and intercostal muscles, at the intersection point of the anterior axillary line and the level of the nipple (at the level of the 4th-5th ribs).
  It has a wide range of use for postoperative pain management in trauma surgery, cardiac surgery, thoracic surgery and breast surgery.
  Other Names: serratus anterior plane block
Procedure: DSAPB — The SAP block, which is among the chest wall blocks, provides its effect by blocking the lateral cutaneous branches of the T2-T9 intercostal nerves, n. intercostobrachial , n. longus thoracicus , n. thoracodorsal.
  SAP block can be performed in two ways: superficial and deep. The deep SAP block is administered between the serratus anterior and intercostal muscles, at the intersection point of the anterior axillary line and the level of the nipple (at the level of the 4th-5th ribs). Following hydrodissection between the serratus anterior and intercostal muscles, a single-shot injection is administered. Subsequently, a peripheral nerve block catheter is placed in the same region under ultrasound guidance.
  Other Names: serratus anterior plane peripheral block cathather replacement
  Arms: DSAPB

SUMMARY:
The aim of this observational study is to compare the analgesic efficacy of continuous infusion via peripheral catheter versus single-shot serratus anterior plane block in women aged 18 to 80 undergoing breast-conserving surgery. The main questions it aims to answer are: Does continuous serratus anterior plane block via peripheral catheter provide superior postoperative analgesic efficacy compared to single-shot serratus anterior plane block? Second question is: Does continuous infusion via catheter in peripheral nerve blocks reduce the amount of intravenous analgesics consumed and improve patient comfort?

ELIGIBILITY:
Inclusion Criteria:

* Female patients aged 18 to 80 years
* Scheduled for breast-conserving surgery
* Classified as American Society of Anesthesiologists (ASA) physical status I, II, or III

Exclusion Criteria:

* Patients with coagulopathy
* Patients with wounds or infections at the block site
* Patients with known allergy to local anesthetic agents
* Patients with mental retardation or limited cooperation
* Patients who do not consent to participate in the study
* Patients who, for any reason, discontinue participation during the course of the study

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2025-01-26 (Actual); Primary Completion 2025-04-26 (Actual); Study Completion 2025-05-26 (Actual)

PRIMARY OUTCOMES:
Numeric Rating Scale | Until discharge after surgery, during an average hospital stay of approximately 24 hours.
  1 - 10
  1 is minimum pain 10 is maximum pain the lower scale is better for pain management.

CONTACTS AND LOCATIONS:
Locations (1):
- Göztepe Prof. Dr. Süleyman Yalçın Şehir Hastanesi, Istanbul, Kadıköy, Turkey (Türkiye)